CLINICAL TRIAL: NCT07200778
Title: Reducing Operative Blood Loss in Laparoscopic Myomectomy With Umbilico-uterine Trunk Clipping
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Mohamed Hassan Mohamed Abdel Ghfar, Lecturer of Obstetrics and Gynecology, Minia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 1531-5-2025
Record Dates: First submitted 2025-09-23; First posted 2025-10-01 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Laparoscopic Myomectomy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): participants will undergo umbilico-uterine trunk occlusion
  Interventions: Procedure: umbilico-uterine trunk occlusion
- Group B (Active Comparator): participants will undergo local injections of epinephrine into the serosal and/or myometrium, covering the myoma before the uterine incision
  Interventions: Procedure: local epinephrine infiltration

INTERVENTIONS:
Procedure: umbilico-uterine trunk occlusion — participants will undergo umbilico-uterine trunk occlusion during laparoscopic myomectomy
  Arms: Group A
Procedure: local epinephrine infiltration — participants will undergo local injections of epinephrine into the serosal and/or myometrium, covering the myoma before the uterine incision during laparoscopic myomectomy
  Arms: Group B

SUMMARY:
the purpose of this study is to examine how Umbilico-uterine trunk occlusion reduces surgery-associated blood loss in Laparoscopic Myomectomy.

ELIGIBILITY:
Inclusion Criteria:

* Age between 19 and 45
* Symptoms of menorrhagia, pelvic pain, or infertility
* Plan to have a laparoscopic myomectomy
* Number of myomas ≤ 4, with the largest myoma measuring ≤ 9 cm

Exclusion Criteria:

* Postmenopausal status
* Dominant pedunculated subserosal FIGO classification (6-7)
* Submucosal type of myoma FIGO classification (0-2)
* Suspicion of malignant uterine or adnexal diseases
* Major medical comorbidities or psychiatric illnesses that could affect follow-up and/or compliance
* Refusal to participate or provide consent to the procedures.

Ages: 19 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 66 (Estimated)
Dates: Start 2025-09-11 (Actual); Primary Completion 2026-03-11 (Estimated); Study Completion 2026-03-11 (Estimated)

PRIMARY OUTCOMES:
Operative Blood Loss | during operation
  The difference between the total amount of irrigation and suction will be used to compute operational blood loss
Hemoglobin drop | 24 hours postoperative
  The difference between the preoperative and postoperative hemoglobin levels will be used to define the hemoglobin change.

CONTACTS AND LOCATIONS:
Locations (1):
- Minia advanced laparoscopy unit, Minya, Egypt